CLINICAL TRIAL: NCT03578991
Title: Diabetes as an Accelerator of Cognitive Impairment and Alzheimer's Disease: Comprehensive Approach and Adherence to Treatment: DIALCAT Project.
Brief Title: Diabetes as an Accelerator of Cognitive Impairment and Alzheimer's Disease
Acronym: DIALCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Sanitari Pere Virgili (Other)
Collaborators: Hospital Vall d'Hebron (Other); Consorci Sanitari de Terrassa (Other); Fundació Recerca Mútua Terrassa (FMT) (Unknown); Clínica Universitària de la Fundació Universitària del Bages (FUB) (Unknown); Althaia Xarxa Assistencial Universitària de Manresa (Other); Fundació Privada Hospital Asil de Granollers (HAG) (Unknown); Consorci Hospitalari de Vic (Other); LambdaLoopers (Other); Universitat Politècnica de Catalunya (Other); Leitat (Unknown); Mixestat (Unknown); Meditecnologia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIALCAT COMRDI-B64574221423350; COMRDI B64574221423350 (Other Grant/Funding Number: Fons Europeu de Desenvolupament Regional (FEDER) & ACCIÓ)
Record Dates: First submitted 2018-06-20; First posted 2018-07-06 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Patients Aged 65-85 (Both Included); Diagnosed of Mild Cognitive Impairment; Diagnosed of Type 2 Diabetes in Active Treatment (Hypoglycemic Agents) for a Period ≥5 Years
Keywords: Type 2 diabetes mellitus; Mild cognitive impairment; Alzheimer disease; Intervention; Clinical trial; mHealth; Smart electronic pillbox; Interactive digital platform
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (No Intervention): Control group - Treatment as usual:
  Type 2 diabetic patients with mild cognitive impairment who will receive the standard clinical treatment recommended by their primary care physician/endocrinologist.
- Arm 2 (Experimental): Intervention - Smart pillbox:
  Type 2 diabetic patients with mild cognitive impairment receiving the standard clinical treatment recommended by their primary care physician/endocrinologist, plus the use of a smart pillbox.
  Interventions: Device: Smart pillbox
- Arm 3 (Experimental): Intervention - Smart pillbox & Interactive digital platform:
  Description: Type 2 diabetic patients with mild cognitive impairment receiving the standard clinical treatment recommended by their primary care physician/endocrinologist, plus the use of a smart pillbox and an interactive digital platform.
  Interventions: Device: Smart pillbox; Other: Interactive digital platform

INTERVENTIONS:
Device: Smart pillbox — The smart electronic pillbox will monitor adherence to pharmacological treatment by means of registering time of medications intake. It will incorporate visual and auditory reminders for taking medications (all of them, being or not being inside the dispenser such as insulin or eye drops). The dispenser will also have sensors and alarms to ensure the proper preservation of the medicines contained. The dispenser will be recharged weekly by a trained pharmacist. Each dispenser will be identified unequivocally with one user, and it will be interconnected with a mobile application (app).
  Arms: Arm 2; Arm 3
Other: Interactive digital platform — The digital interactive platform will allow communication between patients and caregivers and healthcare professionals. Its aims are to provide feedback and guidelines on treatment adherence and also, on how to better optimize treatment on cardiovascular risk factors. The platform will inform about medication dosages and intake schedule, healthy lifestyles related to diabetes, occurrence of adverse events, and it will also monitor patients' glycemic control. In this sense, several alarms are programmed to warn caregivers or even healthcare professionals when the patient has hyperglycemia or hypoglycaemia. The platform will provide too guidelines on how to treat hypo or hyperglycemia as well as most common adverse events, and it will describe reasons to have suffered it.
  Arms: Arm 3

SUMMARY:
This randomized controlled trial is aimed at studying the effects of an eHealth intervention on improving metabolic control and other cardiovascular risk factors (obesity, lipidic profile and hypertension) as the approach to prevent or delay the process of cognitive impairment, and to reduce conversion rates to Alzheimer's disease (AD) in a sample of patients diagnosed of type 2 diabetes mellitus (T2D) and with mild cognitive impairment (MCI).

For these purposes, the standard clinical treatment for this type of patients will be compared with two types of interventions (parallel groups): one aimed at promoting adherence to treatment through the use of a smart pillbox; and the other intervention will be based on the use of the smart pillbox plus and interactive digital platform allowing communication between patients and caregivers with healthcare professionals. Both interventions are targeted to improve adherence to treatment.

The hypothesis is that the rate of conversion from MCI to AD will be higher in the control group than in the intervention groups (higher conversion rates are expected in control group, followed by the smart pillbox group, and lower conversion rates are expected in the group using the interactive digital platform and the smart pillbox).

DETAILED DESCRIPTION:
The objective of the DIALCAT randomized controlled trial is to study the effects of an eHealth intervention (smart pillbox, digital platform) on the progression of cognitive impairment evaluated by means of a neuropsychological examination, in a sample of elderly patients with type II diabetes (T2D) and mild cognitive impairment (MCI). As secondary goals, this research is intended to:

1. Assess if the intervention improves the metabolic control of the study sample.
2. Evaluate the effects of the intervention on the conversion rate (yes vs. no) from MCI to Alzheimer's' disease (AD).
3. Compare the effectiveness of the interventions to reduce functional decline (quantified by a battery of neuropsychological tests [see detailed description below]) and the conversion rate to AD.
4. Identify the clinical and analytical predictors (biomarkers) of conversion from MCI to AD.

To this purposes, a total of 174 T2D patients with MCI (MMSE≥24) will be recruited with a 18-month follow-up. Eligible patients will be randomized in a 1:1:1 ratio in one of the arms of the RCT (for randomization, a sex-by-sex-swapped sequence and the ApoE genotype will be used). The three groups will receive the following interventions:

Arm 1: T2D patients (n = 58) with MCI, receiving treatment as usual (TAU) by their primary care physician/endocrinologist.

Arm 2: T2D patients (n = 58) with MCI, receiving TAU and using a smart pillbox that allows to monitor adherence to treatment.

Arm 3: T2D patients (n = 58) with MCI, receiving TAU, using the smart pillbox and receiving periodic feedback on their metabolic control and how to improve it by an endocrinologist via a digital platform.

Since it is expected that the different factors related to the intervention will have an additive or synergistic effect, the hypothesis is that the cognitive impairment and progression of MCI to AD would be higher in arm 1, followed by arm 2 and, finally, arm 3.

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed of diabetes mellitus type 2 with time evolution ⋝5 years.
2. Age between 65 and 85 years old (both included).
3. Ability to read and write.
4. Active treatment with hypoglycemic agents.
5. Diagnosed with mild cognitive impairment.

Exclusion Criteria:

1. Familiar history of Alzheimer's' disease.
2. Patients with any type of dementia.
3. History of neurological or psychiatric conditions not stabilized that can substantially affect cognition.
4. Severe metabolic or systemic disease that affects the cognitive state. This includes:

   * Unstable acute cardiovascular disease.
   * Renal failure with glomerular filtration rate <30 ml/min/m2.
   * Decompensated cirrhosis or liver failure.
   * Untreated hypothyroidism or vitamin B12 deficiency. If known.
   * Active cancer or chemotherapy treatment the previous year.
5. Treatment with drugs that alter the cognitive state, for example:

   * Antipsychotic.
   * Daily consumption of opioids.
   * Benzodiazepines (BZD) long action (for example Diazepam). Benzodiazepines (BZD) short-acting at high doses such as Alprazolam at doses greater than 1 mg / day; Lorazepam at doses greater than 1 mg / day and Lormetazepam at doses greater than 1 mg / day.
   * Fentanil patches in doses greater than 2.5 mg every 72 h.
   * Gabapentin in doses greater than 600 mg / day.
   * Pregabalin in doses greater than 50 mg / day.
   * Amitriptyline in doses greater than 25 mg / day.
6. Limitations of mobility that can avoid or restrict the application or evaluation of the intervention.
7. Patients with other types of diabetes: diabetic mellitus type 1, LADA; MODY
8. Unstable advanced diabetic retinopathy
9. Patients with serious uncorrected sensory deficits that make assessment impossible (blindness, deafness).
10. Patients with access to other online platforms for patients.
11. Patients with access to other intelligent electronic dispensing devices for improved adherence to treatment.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change of score obtained in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  The main variable of the study will be the score obtained in the RBANS in the different assessment periods. The RBANS was designed to be administered in adult population between 20 and 89 years. It is sensitive to the detection of cognitive disorder in degenerative and non-degenerative pathology. This battery evaluates 5 functions, by means of 12 subtests: 1) attention (repetition of digits and numerical key), 2) language (designation of drawings and semantic fluency), 3) visual-espacial / constructive ability (copy a figure and orientation of lines), 4) immediate memory (word learning and memory of the story) and 5) deferred memory (record of the list, word recognition, record of the story, record of the figure). The RBANS is a short battery (time of administration ≦30 minutes), and has two parallel forms of evaluation (forms A and B) to avoid the effect of learning.

SECONDARY OUTCOMES:
Cardiovascular risk factor: Hypertension. | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  Hypertension (mmHg) will be registered. Both pressures will be assessed (systolic and diastolic). This information will be extracted from clinical records.
Cardiovascular risk factor: Obesity. | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  Body Mass Index (BMI) will be calculated. Weight and height will be combined to calculate and report BMI. This information will be extracted from clinical records.
Cardiovascular risk factor: Dyslipidemia. | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  Dyslipidemia (md/dL) will be screened. This information will be extracted from clinical records.
Degree of diabetes control. | At baseline (at the moment of the study enrollment), at 9 and an average of 18 months after enrollment.
  For the degree of diabetes control will be registered from blood tests level of glycosylated hemoglobin, plasma glucose and insulinemia in fasting.
Usal medication. | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  Medication for hypertension, dyslipidemia and diabetes will be extracted from clinical records. Type of treatment, dosage, route of administration, frequency and changes in medication will be registered and listed.
Presence of micro and macrovascular complications. | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  The presence and severity of retinopathy, nephropathy (microalbuminuria levels), polyneuropathy and/or cardiovascular disease (specifically, ischemic heart disease, cerebrovascular accident or peripheral arterial disease) will be extracted from medical records.
Presence and severity of hypoglycemia. | At baseline (at the moment of the study enrollment), at 4, 9, 13 and an average of 18 months after enrollment.
  Patients will be asked about the presence and severity of hypoglycaemia by answering a self-reported measure developed ad hoc by the Endocrinology Service of the Vall d'Hebron University Hospital. Patients with ambulatory insulinization will have a glucometer which will be reviewed by the doctor at each visit. Wil considerate hypoglycemia when the capillary glucose levels are between 70-50 mg/dl, and hypoglycemia when the levels are <50 mg/dl. All hypoglycemia will be registered.
Lipid profile and renal and hepatic function. | At baseline (at the moment of the study enrollment), at 9 and an average of 18 months after enrollment.
  Levels of low-density lipoprotein cholesterol (mg/dl), high-density lipoprotein cholesterol (mg/dl), triglycerides (mg/dl), creatinine (mg/dl), glomerular filtration (ml/min/m2), aspartate aminotransferase (U/L) and alanine aminotransferase (U/L) will be registered by means of blood tests. A final composite (bad vs. good lipidic profile and hepatic function) will be calculated based on these parameters.
Biomarkers (serum and DNA). | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  Biomarkers (serum and DNA) will be registered by means of blood tests.
Short Physical Performance Battery test (SPPB). | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  The SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Hachinski Scale (HS). | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  The HS allows differentiation of degenerative vascular dementias. A score ≥7 suggests vascular dementia and a score <4 points suggests Alzheimer's disease. The validity of this scale has been investigated in several clinical studies, considering a specificity and sensitivity of the order of 70-80%.
Blessed Dementia Rating Scale (BDRS). | At baseline (at the moment of the study enrollment), at, 4, 9, 13 and an average of 18 months after enrollment.
  The BDRS allows to screen for MCI and dementia in the elderly by quantifying performance in daily life activities by means of 28 items. The sensitivity according to the Cambridge Mental Disorders of the Elderly Examination (CAMCOG) was 90% with a specificity of 76%. A score >15 suggests moderate or severe dementia; a score between 4-14 suggests suspicion of dementia.
Geriatric Depression Scale (GDS; 15-item short form). | At baseline (at the moment of the study enrollment), at, 4, 9, 13 and an average of 18 months after enrollment.
  The Geriatric Depression Scale (GDS) is one of the most widely used instrument for the screening of depression in the elderly. This auto-administered questionnaire have shown to be sensitive to depression among elderly persons suffering from mild to moderate dementia and physical illness. The 15-item short version of the GDS (GDS-15) is considered useful in situations where economy of time is required. The score of the GDS-15 ranges from 0 to 15. A score of zero to four is considered to be within the normal range, five to nine indicates mild depression, and a score of 10 or more indicates moderate to severe depression.
Schwab and England Activities of Daily Living Scale (SE-ADL). | At baseline (at the moment of the study enrollment), at 4, 9, 13 and an average of 18 months after enrollment.
  This scale describing the capacity for daily living shown by a patient with Parkinson's Disease and can be used for other conditions. This scale uses a percentage system to assign levels of independence and dependence, in which 100 percent represents complete independence and 0 percent complete dependence (bedridden).
Montreal Cognitive Assessment (MOCA). | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  The MOCA is a cognitive screening test for MCI and Early Alzheimer's disease. According to the validation study, the sensitivity and specificity of the MOCA for detecting MCI were 90% and 87% respectively. Is a one-page 30-point test administered in approximately 10 minutes.
Mini-Mental State Examination (MMSE). | At baseline (at the moment of the study enrollment), and an average of 18 months after enrollment.
  The MMSE is a brief cognitive test that assesses several cognitive domains, such as orientation, attention, concentration, memory, language, and constructional abilities. For the MMSE the sensitivity was 0.87 and 0.82 for specificity.
Memory failure in everyday life questionnaire (MFE). | At baseline (at the moment of the study enrollment), at 4, 9, 13 and an average of 18 months after enrollment.
  The MFE is one of the most widely-used instruments to assess memory failures in daily life to detect cognitive complaints. It consists of 28 items and has revealed a sensitivity of 83.1% with a specificity of 81.8% and positive predictor vale of 95.3%.
The Functional Social Support Questionnaire (DUKE-UNC-11). | At baseline (at the moment of the study enrollment), at 4, 9, 13 and an average of 18 months after enrollment.
  The DUKE-UNC-11 allows to measure the patient perception of the amount and type of personal social support. It was originally developed to measure social support in family medicine patients. Cut-off lower than 32 indicates low self-perceived social support.
The Resource Utilization in Dementia (RUD). | At baseline (at the moment of the study enrollment), at 9 and an average of 18 months after enrollment.
  The RUD instrument is valid for assessing healthcare resource utilization among older adults with dementia and their caregivers, and time spent on formal and informal care by caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Inzitari, MD, PhD, Principal Investigator — Parc Sanitari Pere Virgili
Locations (8):
- Spain (8):
  - Fundació Privada Hospital Asil de Granollers (HAG), Granollers, Barcelona
  - Fundació Althaia (FA), Manresa, Barcelona
  - Fundació Recerca Mútua Terrassa (FMT), Terrassa, Barcelona
  - Consorci Sanitari de Terrassa (CST), Terrassa, Barcelona
  - Consorci Hospitalari de Vic (CHV), Vic, Barcelona
  - Parc Sanitari Pere Virgili, Barcelona
  - LambdaLoopers, Barcelona
  - University Hospital Vall d'Hebron - Vall d'Hebron Institute of Research, Barcelona

IPD SHARING:
Plan to Share IPD: No